CLINICAL TRIAL: NCT00406653
Title: A Phase 3, Multi-Center, Randomized, Placebo-Controlled Study to Evaluate the Clinical Efficacy and Safety of Induction and Maintenance Therapy With Abatacept in Subjects With Active Crohn's Disease (CD) Who Have Had an Inadequate Clinical Response and/or Intolerance to Medical Therapy
Brief Title: A Study of Abatacept in Patients With Active Crohn's Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IM101-084
Record Dates: First submitted 2006-12-01; First posted 2006-12-04 (Estimated); Results first posted 2010-08-31 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): 4 arms for induction period
  2 arms for maintenance period
  Interventions: Drug: abatacept
- 2 (Placebo Comparator): 4 arms for induction period
  2 arms for maintenance period
  Interventions: Drug: placebo
- abatacept (Other): 1 arm for open-label extension phase
  Interventions: Drug: abatacept

INTERVENTIONS:
Drug: abatacept — Dextrose 5% in water, intravenous (IV).
  Placebo on days Induction Period (IP)-1, IP-15,IP-29, IP-57;
  3 mg/kg on days IP-1, IP-15,IP-29, IP-57;
  ~10 mg/kg on days IP-1, IP-15,IP-29, IP-57,
  or 30 mg/kg on days IP-1,IP-15 and ~10 mg/kg on days IP-29, IP-57.
  Induction Period 3 months
  Maintenance Period 12 months
  Other Names: Orencia; BMS-188667
  Arms: 1
Drug: placebo — Normal saline, IV, 0 mg/kg, every 28 days.
  Induction Period 3 months
  Maintenance Period 12 months
  Arms: 2
Drug: abatacept — ~10 mg/kg, every 28 days.
  Open- Label Extension Period until the drug is marketed for Crohn's Disease (CD)or the CD development program for abatacept is discontinued
  Other Names: Orencia; BMS-188667
  Arms: abatacept

SUMMARY:
The purpose of this clinical research study is to learn if abatacept can improve signs and symptoms of active Crohn's Disease in patients who have not had an adequate response to other therapies. The safety of this treatment will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* have had Crohn's Disease for at least 3 months
* moderate to severely active Crohn's Disease
* have had an inadequate response or intolerance to other Crohn's Disease treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 451 (Actual)
Dates: Start 2006-12; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (100):
- United States (37):
  - University Of Alabama Medical Center, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - The Permanente Medical Group, Inc, Sacramento, California
  - University Of Florida, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Shafran Gasteroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - University Of Chicago Hospitals, Chicago, Illinois
  - Health Science Center, Pratt, Kansas
  - University Of Kentucky Medical Center, Lexington, Kentucky
  - University Of Louisville, Louisville, Kentucky
  - Gulf Coast Research Assoc, Baton Rouge, Louisiana
  - Vanderlick, Michael, Lafayette, Louisiana
  - Maryland Digestive Disease Research, Laurel, Maryland
  - Minnesota Gastroenterology, P.A., Plymouth, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Kansas City Gastroenterology And Hepatology, Kansas City, Missouri
  - Aga Clinical Research Associates, Llc, Egg Harbor Twp, New Jersey
  - Long Island Clinical Research, Great Neck, New York
  - Mount Sinai School Of Medicine, New York, New York
  - U Of Rochester Gastroenterology And Hepatology, Rochester, New York
  - University Endoscopy Center, Syracuse, New York
  - University Of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology & Hepatology, Pllc, Charlotte, North Carolina
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Gastroenterology Specialists, Inc., Canton, Ohio
  - Consultants For Clinical Research, Cincinnati, Ohio
  - Gastrointestinal & Liver Diseases Consultants, Dayton, Ohio
  - Options Health Research, Llc, Tulsa, Oklahoma
  - Allegheny Center For Digestive Health, Pittsburgh, Pennsylvania
  - Southeastern Clinical Research, Chattanooga, Tennessee
  - Gastroenterology Center Of The Midsouth, P.C., Germantown, Tennessee
  - Memphis Gastroenterology Group, Germantown, Tennessee
  - Nashville Medical Research, Nashville, Tennessee
  - Austin Gastroenterology, Pa, Austin, Texas
  - Gastroenterology Clinic Of San Antonio, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Australia (10):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Herston, Queensland
  - Local Institution, South Brisbane, Queensland
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Launceston, Tasmania
  - Local Institution, Box Hill, Victoria
  - Local Institution, Fitzroy, Victoria
  - Local Institution, South Ballarat, Victoria
  - Local Institution, Fremantle, Western Australia
- Belgium (3):
  - Local Institution, Bonheiden
  - Local Institution, Leuven
  - Local Institution, Roeselare
- Brazil (5):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Goiânia, Goiás
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
- Canada (9):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Halifax, Nova Scotia
  - Local Institution, London, Ontario
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
- Local Institution, České Budějovice, Czechia
- Denmark (4):
  - Local Institution, Aalborg
  - Local Institution, Arhus C
  - Local Institution, Hvidovre
  - Local Institution, Odense C
- France (6):
  - Local Institution, Amiens
  - Local Institution, Lille
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac
  - Local Institution, Toulouse
- Germany (2):
  - Local Institution, Kiel
  - Local Institution, Münster
- India (6):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Hyderabad
  - Local Institution, Mangalore
  - Local Institution, Manipal
  - Local Institution, Mumbai
  - Local Institution, Mysore
- Italy (4):
  - Local Institution, Napoli
  - Local Institution, Padua
  - Local Institution, Roma
  - Local Institution, San Giovanni Rotondo
- Mexico (3):
  - Local Institution, Torreón, Coahuila
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
- Netherlands (3):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Rotterdam
- Local Institution, Katowice, Poland
- Local Institution, Ponce, Puerto Rico
- South Africa (2):
  - Local Institution, Overport, KwaZulu-Natal
  - Local Institution, Belville, Western Cape
- Switzerland (3):
  - Local Institution, Bern
  - Local Institution, Lausanne
  - Local Institution, Zurich

REFERENCES:
- [Derived] Sandborn WJ, Colombel JF, Sands BE, Rutgeerts P, Targan SR, Panaccione R, Bressler B, Geboes K, Schreiber S, Aranda R, Gujrathi S, Luo A, Peng Y, Salter-Cid L, Hanauer SB. Abatacept for Crohn's disease and ulcerative colitis. Gastroenterology. 2012 Jul;143(1):62-69.e4. doi: 10.1053/j.gastro.2012.04.010. Epub 2012 Apr 12. PMID 22504093

RESULTS

PARTICIPANT FLOW:
Groups:
- Abatacept (ABA) 30/~10 mg/kg, Induction Period (IP): During IP, abatacept administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (10 mg/kg group).
- ABA ~10 mg/kg, IP: During IP, abatacept administered IV on Days IP-1, IP-15, IP-29, and IP-57 at a dose of ~10 mg/kg (weight-tiered).
- ABA 3 mg/kg, IP: During IP, abatacept administered IV on Days IP-1, IP-15, IP-29, and IP-57 at a dose of 3 mg/kg (fixed dose).
- Placebo, IP: During the IP, placebo was administered IV on Days IP-1, IP-15, IP-29, and IP-57.
- ABA ~10 mg/kg, Maintenance Period (MP): During MP, abatacept administered IV at a dose of ~10 mg/kg (weight-tiered dosing) every 28 days starting Day MP-1.
- Placebo, MP: During MP, placebo was administered IV at 28-day intervals starting on Day MP-1.
- ABA ~10 mg/kg, Open-Label Period (OL): During OL, abatacept administered IV at a dose of ~10 mg/kg (weight-tiered dosing) every 28 days starting Day OL-1.
Period: Induction Period
Arm/Group | Abatacept (ABA) 30/~10 mg/kg, Induction Period (IP) | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP | ABA ~10 mg/kg, Maintenance Period (MP) | Placebo, MP | ABA ~10 mg/kg, Open-Label Period (OL)
Started | 65 | 128 | 130 | 128 | 0 | 0 | 0
Completed | 50 | 94 | 112 | 102 | 0 | 0 | 0
Not Completed | 15 | 34 | 18 | 26 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 10 | 4 | 11 | 0 | 0 | 0
Not completed — Lack of Efficacy | 11 | 14 | 8 | 10 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal of Consent | 2 | 5 | 1 | 2 | 0 | 0 | 0
Not completed — Subject No Longer Meets Study Criteria | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Declined participation but followup done | 0 | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Given prohibited drug | 0 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Incarcerated | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Patient relocated | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | Abatacept (ABA) 30/~10 mg/kg, Induction Period (IP) | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP | ABA ~10 mg/kg, Maintenance Period (MP) | Placebo, MP | ABA ~10 mg/kg, Open-Label Period (OL)
Started | 0 | 0 | 0 | 0 | 44 (At end of IP, 44 participants met response criteria and were randomly assigned to abatacept in MP.) | 46 (At end of IP, 46 participants met response criteria and were randomly assigned to placebo in MP.) | 0
Completed | 0 | 0 | 0 | 0 | 14 | 10 | 0
Not Completed | 0 | 0 | 0 | 0 | 30 | 36 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 20 | 26 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Administrative Reason By Sponsor | 0 | 0 | 0 | 0 | 4 | 7 | 0
Not completed — Error in disease score evaluation | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Open-Label Period
Arm/Group | Abatacept (ABA) 30/~10 mg/kg, Induction Period (IP) | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP | ABA ~10 mg/kg, Maintenance Period (MP) | Placebo, MP | ABA ~10 mg/kg, Open-Label Period (OL)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 324 (All completing IP but failing response criteria and those completing or relapsing on MP entered OL.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 324
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 18
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 160
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Withdrawal of Consent | 0 | 0 | 0 | 0 | 0 | 0 | 11
Not completed — Subject No Longer Meets Study Criteria | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Administrative Reason By Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 115
Not completed — Declined participation but followup done | 0 | 0 | 0 | 0 | 0 | 0 | 8
Not completed — Discontinued by Sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Refused followup | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ABA 30/~10 mg/kg, Induction Period (IP): During IP, abatacept administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (10 mg/kg group).
- Total: Total of all reporting groups
Arm/Group | ABA 30/~10 mg/kg, Induction Period (IP) | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP | Total
Number analyzed (Participants) | 65 | 128 | 130 | 128 | 451
Age Continuous [Mean (Standard Deviation); unit: years] | 36.0 (11.12) | 38.6 (12.90) | 36.9 (13.35) | 38.0 (12.98) | 37.6 (12.81)
Age, Customized [Number; unit: Participants]
  <30 years | 23 | 37 | 51 | 41 | 152
  Between 30 and 50 years | 35 | 64 | 57 | 64 | 220
  >50 years | 7 | 27 | 22 | 23 | 79
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 78 | 78 | 83 | 277
  Male | 27 | 50 | 52 | 45 | 174
Region of Enrollment [Number; unit: participants]
  United States | 24 | 45 | 46 | 38 | 153
  Italy | 0 | 5 | 5 | 5 | 15
  Switzerland | 2 | 4 | 3 | 1 | 10
  India | 1 | 3 | 2 | 2 | 8
  France | 6 | 8 | 7 | 7 | 28
  Czech Republic | 1 | 2 | 0 | 2 | 5
  Mexico | 1 | 4 | 0 | 3 | 8
  Puerto Rico | 1 | 0 | 0 | 2 | 3
  Canada | 8 | 18 | 22 | 27 | 75
  Brazil | 3 | 7 | 6 | 6 | 22
  Belgium | 2 | 7 | 9 | 13 | 31
  Korea, Democratic People's Republic of | 1 | 1 | 1 | 1 | 4
  Denmark | 1 | 4 | 10 | 2 | 17
  Australia | 6 | 10 | 13 | 13 | 42
  South Africa | 5 | 5 | 1 | 2 | 13
  Germany | 0 | 2 | 2 | 3 | 7
  Netherlands | 3 | 3 | 3 | 1 | 10
Inadequate Response/Intolerance to Prior Anti-Tumor Necrosis Factor (TNF) Agent Therapy [Number; unit: Participants] — Prior to this study, participants had an inadequate response and/or intolerance to an approved anti-tumor necrosis factor (TNF) agent at an approved labeled dose for at least 8 weeks.
  Participants
    Inadequate Response/Intolerance To Prior Agents | 42 | 86 | 77 | 77 | 282
    No Inadequate Response/Intolerance To Prior Agents | 23 | 42 | 53 | 51 | 169
Crohn's Disease (CD) Duration [Mean (Standard Deviation); unit: Years] — Clinical diagnosis of CD with active disease confirmed by endoscopic, histologic, or radiographic evidence using established diagnostic criteria.
  Years | 8.4 (7.49) | 9.9 (8.74) | 9.2 (7.98) | 9.8 (8.29) | 9.5 (8.21)
Crohn's Disease Activity Index (CDAI) [Mean (Standard Deviation); unit: points] — CDAI is a composite index consisting of a weighted scoring of 8 disease variables: number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI scores range from 0 to ~600 points. Clinical response=CDAI reduction ≥100 points or absolute CDAI <150 points. Clinical remission=CDAI <150 points. Moderate to severe disease=CDAI ≥220 and ≤450 points.
  points | 320.6 (61.59) | 318.9 (65.08) | 317.9 (59.87) | 320.7 (72.09) | 319.4 (65.03)
Inflammatory Bowel Disease Questionnaire (IBDQ) Score [Mean (Standard Deviation); unit: units on a scale] — IBDQ was used to measure disease specific quality of life. The IBDQ consists of a self-administered 32-item questionnaire that evaluates quality of life across 4 dimensional scores: Bowel, Systemic, Social and Emotional. The response to each question can range from 1 to 7, with 1 indicating severe problem and 7 indicating normal health. The total IBDQ is computed as the sum of the responses to the individual IBDQ questions. The total score can range between 32 to 224 with higher scores indicating a better quality of life.
  units on a scale | 119.9 (26.22) | 117.3 (30.60) | 121.1 (28.0) | 119.6 (31.17) | 119.5 (29.36)

OUTCOME MEASURES:

1. Primary Outcome: Induction Period (IP); Number of Participants With Crohn's Disease Activity Index (CDAI)-Defined Clinical Response at Both Day IP-57 and Day IP-85
Description: CDAI is a composite index consisting of a weighted scoring of 8 disease variables:number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score was based partly on entries (7 days before evaluation) from participant's Diary kept while on study. CDAI scores range from 0 to ~600 points. Clinical response=CDAI reduction ≥100 points or absolute CDAI <150 points. Clinical remission=CDAI <150 points. Moderate to severe disease=CDAI ≥220 and ≤450 points.
Time Frame: At both Day IP-57 (Wk 8) and Day IP-85 (Wk 12).
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Induction Period. Due to site non-compliance with the study protocol, 1 randomized and treated participant from Site 166 was excluded.
Measure: Number; unit: participants
Groups:
- ABA 30/~10 mg/kg, IP: During IP, abatacept administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (10 mg/kg group).
- ABA ~10 mg/kg, IP: During IP, abatacept administered IV on Days IP-1 and IP-15 at a dose of ~10 mg/kg (weight-tiered). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (weight-tiered; ~10 mg/kg group).
- ABA 3 mg/kg, IP: During IP, abatacept administered IV on Days IP-1 and IP-15 at a dose of 3 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of 3 mg/kg (3 mg/kg group).
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 64 | 128 | 129 | 125
participants | 11 | 13 | 20 | 18
Statistical Analysis 1: Comparison: ABA 30/~10 mg/kg, IP vs Placebo, IP; Conditional on abatacept (ABA) 30/~10 mg/kg vs placebo (PLA)comparison being statistically significant at 5% significance level, ABA ~10 mg/kg vs PLA to be tested at 5% significance level. Null hypothesis=no treatment difference (relative risk [RR] of ABA over placebo=1).First comparison: power=99%,sample size=134,expected PLA response rate=25%, ABA 30/~10 mg/kg=55%. Cochran-Mantel-Haenszel Chi square p-value and RR along with 95% confidence interval provided, adjusting for randomization strata; Test type: Superiority or Other; p = 0.611, Cochran-Mantel-Haenszel — Due to randomization misspecification, 2:2:2:1 ratio applied instead of planned 2:1:2:2 (placebo, ABA 3mg/kg, ~10mg/kg, 30/~10mg/kg). Only ~half intended number assigned to ABA 30/~10 mg/kg arm and ~double intended number assigned to ABA 3 mg/kg arm; Second primary comparison (conditional on first): power=91%, sample size=134, 5% significance; expected PLA response rate= 25%, ABA/~10 mg/kg=45%; Risk Ratio (RR) = 1.2, 95% CI 2-sided [0.6 to 2.4] — All participants who prematurely discontinued for any reason considered not to have achieved clinical response. Normal approximation used if number of responses in treatment group was ≥5. Otherwise an exact method was used

2. Primary Outcome: Maintenance Period (MP); Number of Participants In CDAI-Defined Clinical Remission (CDAI <150) at Day MP-365 (12 Months)
Description: as for outcome 1
Time Frame: Day MP-365 (12 months) of maintenance therapy
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Maintenance Period. The Maintenance Period was not sized based on power considerations, and thus, no formal statistical hypothesis testing was performed.
Measure: Number; unit: participants
Groups:
- ABA ~10 mg/kg, MP: During MP, abatacept administered IV at a dose of ~10 mg/kg (weight-tiered dosing) every 28 days starting Day MP-1.
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 42 | 45
participants | 10 | 5

3. Primary Outcome: Open-Label Extension Period (OL); Number of Participants With Adverse Events (AEs), Related AEs, Deaths, Serious AEs (SAEs), Related SAEs, and Discontinuation Due to AEs
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. Related AE=relationship of certain, probable, possible, or missing. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: Between Day OL-1 and Day OL-617
Population: All participants who received at least 1 infusion of open-label study medication at any time, based on a participant's received treatment (As Treated Analysis Population). The OL was not sized based on power considerations.
Measure: Number; unit: participants
Groups:
- ABA ~10 mg/kg, OL: During OL, abatacept administered IV at a dose of ~10 mg/kg (weight-tiered dosing) every 28 days starting Day OL-1.
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 324
participants
  AEs | 267
  Related AEs | 128
  Deaths | 1
  SAEs | 86
  Related SAEs | 21
  Discontinuation due to AE | 16

4. Secondary Outcome: IP; Number of Participants in CDAI-defined Clinical Remission at Both Day IP-57 and Day IP-85 (Key Secondary Outcome)
Description: as for outcome 1
Time Frame: At both Day IP-57 (Wk 8) and Day IP-85 (Wk 12) of induction therapy
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Induction Period
Measure: Number; unit: participants
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 64 | 128 | 129 | 126
participants | 5 | 5 | 6 | 8
Statistical Analysis 1: Comparison: ABA 30/~10 mg/kg, IP vs Placebo, IP; Conditional on abatacept (ABA) 30/~10 mg/kg vs placebo (PLA)comparison being statistically significant at 5% significance level, ABA ~10 mg/kg vs PLA to be tested at 5% signficance level. Null hypothesis=no treatment difference (relative risk [RR] of ABA over placebo=1).First comparison: power=95%,sample size=134,expected PLA response rate=15%, ABA 30/~10 mg/kg=35%. Cochran-Mantel-Haenszel Chi square p-value and RR along with 95% confidence interval provided, adjusting for randomization strata; Test type: Superiority or Other; Cochran-Mantel-Haenszel — Due to randomization misspecification, 2:2:2:1 ratio applied instead of planned 2:1:2:2 (placebo, ABA mg/kg, ~10 mg/kg, 30/~10 mg/kg). Only ~half intended number assigned to ABA 30/~10 mg/kg arm and ~double intended number assigned to ABA 3 mg/kg arm; Second primary comparison (conditional on first): power=80%, sample size=134, 5% significance; expected PLA response rate= 15%, ABA/~10 mg/kg=30%; Risk Ratio (RR) = 1.18, 95% CI 2-sided [0.4 to 3.44] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: IP; Number of Participants With CDAI-Defined Clinical Response at Both Day IP-57 and Day IP-85 Analyzed by Cochran-Armitage Trend Test for Dose-Response Relationship
Description: as for outcome 1
Time Frame: At both Day IP-57 (Wk 8) and Day IP-85 (Wk 12) of induction therapy
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Induction Period
Measure: Number; unit: participants
Arm/Group | Placebo, IP | ABA 3 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 30/~10 mg/kg, IP
Number analyzed (Participants) | 125 | 129 | 128 | 64
participants | 18 | 20 | 13 | 11
Statistical Analysis 1: Comparison: Placebo, IP vs ABA 3 mg/kg, IP vs ABA ~10 mg/kg, IP vs ABA 30/~10 mg/kg, IP; The Cochran-Armitage trend test was performed to evaluate whether a relationship existed between the response and dose regimen by comparing the proportion of participants in response across all four treatment arms. Normal approximation was used if the number of responses in a treatment group is at least 5. Otherwise an exact method was used; Test type: Superiority or Other; p = 0.436, Cochran-Armitage Trend Test — All statistical testing was performed at a pre-specified alpha-level of 5%

6. Secondary Outcome: IP; Change From Baseline to Day IP-85 In Inflammatory Bowel Disease Questionnaire (IBDQ)
Description: The Inflammatory Bowel Disease Questionnaire (IBDQ) consists of a self-administered 32-item questionnaire evaluating quality of life across 4 dimensional scores: Bowel, Systemic, Social and Emotional. Responses to each question can range from 1 to 7, with 1 indicating severe problem and 7 indicating normal health. The total IBDQ is computed as the sum of the responses to the individual IBDQ questions. The total score ranges between 32 to 224 with higher scores indicating a better quality of life. Change from Baseline= post-Baseline - Baseline value.
Time Frame: Baseline, Day IP-85
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Induction Period with both Baseline and post-Baseline measurements.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 60 | 116 | 124 | 121
units on a scale | 0.79 (3.974) | 11.10 (2.858) | 7.53 (2.765) | 13.4 (2.798)

7. Secondary Outcome: IP; Number of Participants With Adverse Events (AEs), Related AEs, Deaths, Serious AEs (SAEs), Related SAEs, and Discontinuation Due to AEs
Description: as for outcome 3
Time Frame: Day IP-1 through Day IP-85
Population: All participants who received at least 1 infusion of study medication during the Induction Period, based on a participant's received treatment (As Treated Analysis Population)
Measure: Number; unit: Participants
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 65 | 128 | 130 | 128
Participants
  AEs | 49 | 97 | 96 | 95
  Related AEs | 24 | 47 | 46 | 40
  Deaths | 0 | 0 | 0 | 0
  SAEs | 11 | 22 | 20 | 20
  Related SAEs | 2 | 7 | 9 | 6
  Discontinuation due to AE | 1 | 11 | 5 | 12

8. Secondary Outcome: IP; Number of Participants With Adverse Events (AEs) of Special Interest
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. AEs of special interest are those AEs that may be associated with the use of immunomodulatory drugs, including all infections, serious infections, and opportunistic infections; autoimmune disorders; neoplasms; acute infusional AEs (pre-specified AEs occurring within 1 hour of start of infusion) and peri-infusional AEs (pre-specified AEs occurring within 24 hours of the start of infusion).
Time Frame: Day IP-1 through Day IP-85
Population: All participants who received at least 1 infusion of study medication during the IP, based on a participant's received treatment (As Treated Analysis Population)
Measure: Number; unit: participants
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 65 | 128 | 130 | 128
participants
  All Infections | 13 | 33 | 31 | 42
  Serious Infections | 2 | 9 | 4 | 3
  Opportunistic Infections | 0 | 0 | 0 | 0
  Malignancies-Total | 0 | 0 | 3 | 0
  Malignancies-squamous cell carcinoma | 0 | 0 | 2 | 0
  Malignancies-breast cancer | 0 | 0 | 1 | 0
  Autoimmune Disorders-Total | 2 | 1 | 2 | 2
  Autoimmune Disorders-erythema | 2 | 1 | 2 | 1
  Autoimmune Disorders-psoriasis | 0 | 0 | 0 | 1
  Acute Infusional AEs | 3 | 3 | 4 | 5
  Peri-infusional AEs | 13 | 22 | 15 | 16

9. Secondary Outcome: IP; Number of Participants With Positive Antibody Response to Abatacept (ABA)
Description: A electrochemiluminescent immunoassay screened sera for drug-specific antibodies, immunocompetition identified specific anti-ABA reactivity. Cytotoxic T-Lymphocyte Antigen 4 (CTLA4) and Possibly immunoglobulin (Ig) category= reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity was defined as a post-baseline titer higher than Baseline, or any post-baseline positivity if Baseline value was missing.
Time Frame: For participants treated in MP: Day IP-1 (Baseline) to Day MP-1 (Day IP-85); For participants treated in OL directly after IP: Day IP-1 to Day OL-1; For participants treated only in IP: All measurements after Day IP-1 (including follow-up visits)
Population: All participants who received abatacept and for whom baseline and at least 1 additional measurement were available were included in the Immunogenicity Analysis Population.
Measure: Number; unit: participants
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP
Number analyzed (Participants) | 63 | 123 | 127
participants
  Total | 4 | 7 | 12
  CTLA4/Possibly Ig | 1 | 0 | 6
  Ig and/or Ig Junction | 3 | 7 | 6

10. Secondary Outcome: IP; Number of Participants With CDAI-Defined Clinical Response at Both Day IP-57 and Day IP-85 Among Participants With Inadequate Response and/or Intolerance to Anti-Tumor Necrosis Factor (TNF)
Description: as for outcome 1
Time Frame: At both Day IP-57 (Wk 8) and Day IP-85 (Wk 12) of induction therapy
Population: Participants in the All Randomized and Treated (receiving ≥1 infusion) Population who in the past had an inadequate response to, or who were intolerant to, an approved anti-TNF agent at an approved labeled dose for at least 8 weeks. Due to site non-compliance with the study protocol, 1 randomized and treated participant from Site 166 was excluded.
Measure: Number; unit: participants
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 42 | 86 | 76 | 77
participants | 9 | 8 | 2 | 10

11. Secondary Outcome: IP; Number of Participants in CDAI-Defined Clinical Remission at Both Day IP-57 and Day IP-85 Among Participants With Inadequate Response and/or Intolerance to Anti-TNF
Description: as for outcome 1
Time Frame: At both Day IP-57 (Wk 8) and Day IP-85 (Wk 12) of induction therapy
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | ABA 30/~10 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 3 mg/kg, IP | Placebo, IP
Number analyzed (Participants) | 42 | 86 | 76 | 77
participants | 3 | 2 | 0 | 3

12. Secondary Outcome: IP; Number of Participants Who Are Anti-TNF-Inadequate Responders/Anti-TNF Intolerant With CDAI-Defined Clinical Response at Both Day IP-57 and Day IP-85 Analyzed by Cochran-Armitage Trend Test for Dose-Response Relationship
Description: as for outcome 1
Time Frame: At both Day IP-57 (Wk 8) and Day IP-85 (Wk 12) of induction therapy
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Placebo, IP | ABA 3 mg/kg, IP | ABA ~10 mg/kg, IP | ABA 30/~10 mg/kg, IP
Number analyzed (Participants) | 77 | 76 | 86 | 42
participants | 10 | 2 | 8 | 9
Statistical Analysis 1: Comparison: Placebo, IP vs ABA 3 mg/kg, IP vs ABA ~10 mg/kg, IP vs ABA 30/~10 mg/kg, IP; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.112, Cochran-Armitage Trend Test — All statistical testing was performed at a pre-specified alpha-level of 5%

13. Secondary Outcome: MP; Number of Participants With Adverse Events (AEs), Related AEs, Deaths, Serious AEs (SAEs), Related SAEs, and Discontinuation Due To AEs
Description: as for outcome 3
Time Frame: Between Day IP-85 and Day MP-365
Population: All participants who received at least 1 infusion of study medication during the Maintenance Period, based on a participant's received treatment (As Treated Analysis Population)
Measure: Number; unit: Participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 44 | 46
Participants
  AEs | 31 | 32
  Related AEs | 12 | 15
  Deaths | 0 | 0
  SAEs | 5 | 9
  Related SAEs | 0 | 1
  Discontinuation due to AE | 1 | 0

14. Secondary Outcome: MP; Number of Participants With Adverse Events (AEs) of Special Interest:
Description: as for outcome 8
Time Frame: Between Day IP-85 and Day MP-365
Population: All participants who received at least 1 infusion of study medication during the MP, based on a participant's received treatment (As Treated Analysis Population)
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 44 | 46
participants
  All Infections | 16 | 18
  Serious Infections | 1 | 1
  Opportunistic Infections | 0 | 0
  Malignancies | 0 | 0
  Autoimmune Disorders-Total | 2 | 1
  Autoimmune Disorders-psoriasis | 2 | 0
  Autoimmune Disorders-erythema | 0 | 1
  Acute Infusional AEs | 1 | 0
  Peri-infusional AEs | 2 | 0

15. Secondary Outcome: MP; Number of Participants With Positive Antibody Response to Abatacept
Description: A electrochemiluminescent immunoassay screened sera for drug-specific antibodies, immunocompetition was used to identify specific anti-Abatacept reactivity. CTLA4 and Possibly Ig category= reactivity against extracellular domain of human CTLA4, constant regions of human IgG1, or both (CTLA4Ig; Abatacept molecule). Ig and/or Junction category=reactivity against constant regions and/or hinge region of human IgG1. Drug-induced seropositivity was defined as a post-baseline titer higher than Baseline, or any post-baseline positivity if Baseline value was missing.
Time Frame: For participants not entering OL: All measurements after Day MP-1 (including follow-up visits); For participants entering OL: From first measurement after Day MP-1 to Day MP-365 (Day OL-1)
Population: All participants who received abatacept and for whom baseline and at least 1 additional measurement were available were included in the Immunogenicity Analysis Population. The placebo group was constituted by participants who received abatacept in the IP and underwent drug withdrawal in the MP.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 44 | 40
participants
  Total | 7 | 14
  CTLA4/Possibly Ig | 2 | 8
  Ig and/or Ig Junction | 5 | 8

16. Secondary Outcome: MP; Number of Participants With CDAI-defined Clinical Response at Day MP-365.
Description: as for outcome 1
Time Frame: Day MP-365
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Maintenance Period. Due to site non-compliance with the study protocol, 1 randomized and treated participant from Site 166 was excluded.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 42 | 45
participants | 11 | 7

17. Primary Outcome: OL; Number of Participants With Adverse Events (AEs) of Special Interest
Description: as for outcome 8
Time Frame: Between Day OL-1 and Day OL-617
Population: All participants who received at least 1 infusion of open-label study medication at any time, based on a participant's received treatment (As Treated Analysis Population)
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 324
participants
  All Infections | 144
  Serious Infections | 13
  Opportunistic Infections (OI)-Total | 2
  OI-oral candidiasis | 1
  OI-gastroenteritis Cryptosporidial | 1
  Malignancies-Total | 5
  Malignancies-basal cell carcinoma | 2
  Malignancies-breast cancer | 1
  Malignancies-squamous cell carcinoma | 1
  Malignancies-chronic lymphocytic leukemia | 1
  Autoimmune Disorders-Total | 11
  Autoimmune Disorders-erythema nodosum | 7
  Autoimmune Disorders-psoriasis | 1
  Autoimmune Disorders-pernicious anemia | 1
  Autoimmune Disorders-antiphospholipid syndrome | 1
  Autoimmune Disorders-ankylosing spondylitis | 1
  Acute Infusional AEs | 10
  Peri-infusional AEs | 24

18. Secondary Outcome: MP; Number of Participants in CDAI-defined Clinical Remission at Both Day MP-169 and Day MP-365
Description: as for outcome 1
Time Frame: Day MP-169
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis for the cohort of participants with clinical remission at both Day MP-169 and Day MP-365 was not conducted for the MP as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: MP; Change From Baseline to Day MP-365 in Short Form-36 (SF-36)
Description: The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health; (2) mental component summary=vitality, social functioning, role-emotional, and mental health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: Baseline, Day MP-365
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis for changes from baseline in SF-36 responses were not conducted for the MP as planned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: MP; Change From Baseline to Day MP-365 in Inflammatory Bowel Disease Questionnaire (IBDQ)
Description: as for outcome 6
Time Frame: Baseline, Day MP-365
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis for changes from baseline in IBDQ responses were not conducted for the MP as planned.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

21. Secondary Outcome: MP; Number of Participants Who Were Not On Background Corticosteroid Therapy at Day MP-365 Among All Participants Who Received Baseline Corticosteroid Therapy
Description: Participants who received corticosteroid therapy (e.g. prednisone or budesonide) were to maintain a stable dose until Day MP-1. On or after Day MP-1, a recommended tapering regimen of corticosteroid therapy was planned if the participant was in remission (i.e., CDAI score < 150), or if the participant's condition had satisfactorily improved according to investigators clinical assessment. Other CD therapy was to remain at a stable dose throughout the Maintenance Period, with the exception of decreases due to drug-related toxicities.
Time Frame: Day MP-365
Population: On/after Day MP-1, a recommended tapering of corticosteroids was planned if participant was in remission/had improved. Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analyses for corticosteroid sparing were not conducted for the MP as planned
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: MP; Number of Participants Who Were Not On Background Corticosteroid Therapy at Day MP-365 Among Participants Who Received Baseline Corticosteroid Therapy and Who Achieved CDAI-Defined Clinical Remission
Description: CDAI is a composite index consisting of a weighted scoring of 8 disease variables:number of liquid stools, extent of abdominal pain, general well-being, occurrence of extraintestinal symptoms, need for antidiarrheal drugs, presence of abdominal masses, hematocrit, and body weight. CDAI score is based partly on entries from participant's Diary (7 days before evaluation) which is kept while on study. CDAI scores range from 0 to ~600. Clinical response=CDAI reduction ≥100 or absolute CDAI <150. Clinical remission=CDAI <150. Moderate to severe disease=CDAI ≥220 and ≤450.
Time Frame: Day MP-365
Population: On/after Day MP-1, a defined tapering of corticosteroids was planned if the participant was in remission/had improved. Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analyses for corticosteroid sparing were not conducted for the MP as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

23. Secondary Outcome: MP; Number of Participants With CDAI-Defined Clinical Response Among Participants With Inadequate Response and/or Intolerance to Anti-Tumor Necrosis Factor (TNF)
Description: as for outcome 1
Time Frame: Day MP-365
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint subgroup analysis of clinical response in participants who have had an inadequate response and/or intolerance to anti-TNF therapy was not conducted for the MP as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

24. Secondary Outcome: MP; Number of Participants in CDAI-Defined Clinical Remission Among Participants With Inadequate Response and/or Intolerance to Anti-TNF
Description: as for outcome 1
Time Frame: Day MP-365
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint subgroup analysis of clinical remission in participants who have had an inadequate response and/or intolerance to anti-TNF therapy was not conducted for the MP as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, MP | Placebo, MP
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: OL; Number of Participants Who Were Not On Background Corticosteroid Therapy Among All Participants Who Received Baseline Corticosteroid Therapy
Description: Background corticosteroid therapy included prednisone or budesonide.
Time Frame: Between Day OL-1 and Day OL-617
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis of corticosteroid use in participants was not conducted for the OL as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 0

26. Secondary Outcome: OL; Number of Participants With CDAI-defined Clinical Response or Clinical Remission at Day OL-169
Description: as for outcome 1
Time Frame: Day OL-169
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Open-Label Extension Period.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 163
participants
  Clinical Response | 84
  Clinical Remission | 55

27. Secondary Outcome: OL; Number of Participants With CDAI-defined Clinical Response or Clinical Remission at Day OL-365
Description: as for outcome 1
Time Frame: Day OL-365
Population: All Randomized and Treated (receiving ≥1 infusion) Participants in Open-Label Extension Period.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 69
participants
  Clinical Response | 35
  Clinical Remission | 24

28. Secondary Outcome: OL; Number of Participants With Positive Antibody Response to Abatacept
Description: as for outcome 15
Time Frame: For participants receiving OL medication, all measurements starting after Day OL-1 (including follow-up visits and at 56 and 85 days after last dose)
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 314
participants
  Total | 71
  CTLA4/Possibly Ig | 46
  Ig and/or Ig Junction | 29

29. Secondary Outcome: OL; Number of Participants With Pharmacogenomic Marker Activity
Description: Changes in the expression of individual ribonucleic acid (RNA) transcripts were to be evaluated from whole blood using both microarray transcriptional profiling and quantitative polymerase chain reaction (PCR) methods. Peripheral RNA transcriptional profiling was to be used only to identify individual RNA transcripts that differ in expression with respect to time, treatment and outcome.
Time Frame: Between Day OL-1 and Day OL-617
Population: Due to the early termination of the study after the IP results were reviewed and the primary efficacy endpoint was not achieved, the secondary endpoint analysis of pharmacogenomic marker activity in participants was not conducted for the OL as planned.
Measure: Number; unit: participants
Arm/Group | ABA ~10 mg/kg, OL
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- ABA 30/~10mg/kg (IP): During IP, abatacept administered intravenously (IV) on Days IP-1 and IP-15 at a dose of 30 mg/kg (fixed dose). On Days IP-29 and IP-57, abatacept was administered IV at a dose of ~10 mg/kg (10 mg/kg group).
- ABA 3mg/kg (IP): During IP, abatacept administered IV on Days IP-1, IP-15, IP-29, and IP-57 at a dose of 3 mg/kg (fixed dose).
- ABA ~10mg/kg (IP): During IP, abatacept administered IV on Days IP-1, IP-15, IP-29, and IP-57 at a dose of ~10 mg/kg (weight-tiered).
- ABA ~10mg/kg (MP): During MP, abatacept administered IV at a dose of ~10 mg/kg (weight-tiered dosing) every 28 days starting Day MP-1.
- ABA ~10mg/kg (OL): During OL, abatacept administered IV at a dose of ~10 mg/kg (weight-tiered dosing) every 28 days starting Day OL-1.
- Placebo (IP): During the IP, placebo was administered IV on Days IP-1, IP-15, IP-29, and IP-57.
- Placebo (MP): During MP, placebo was administered IV at 28-day intervals starting on Day MP-1.
Arm/Group | ABA 30/~10mg/kg (IP) | ABA 3mg/kg (IP) | ABA ~10mg/kg (IP) | ABA ~10mg/kg (MP) | ABA ~10mg/kg (OL) | Placebo (IP) | Placebo (MP)
Serious Adverse Events (participants affected / at risk) | 11/65 | 20/130 | 22/128 | 5/44 | 86/324 | 20/128 | 9/46
Other Adverse Events (participants affected / at risk) | 34/65 | 48/130 | 45/128 | 19/44 | 150/324 | 60/128 | 17/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABA 30/~10mg/kg (IP) (N=65) | ABA 3mg/kg (IP) (N=130) | ABA ~10mg/kg (IP) (N=128) | ABA ~10mg/kg (MP) (N=44) | ABA ~10mg/kg (OL) (N=324) | Placebo (IP) (N=128) | Placebo (MP) (N=46)
EPISCLERITIS (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SINUS TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
EMBOLISM (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 2 | 0 | 1 | 1 | 0
ANXIETY (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MAJOR DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
TYPE I HYPERSENSITIVITY (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANTIPHOSPHOLIPID SYNDROME (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
COMPLEX REGIONAL PAIN SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SUBILEUS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
PROCTALGIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
ACUTE ABDOMEN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 3 | 0 | 0
ILEAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CROHN'S DISEASE (Gastrointestinal disorders) | 5 | 9 | 9 | 2 | 35 | 10 | 3
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
SMALL INTESTINAL STENOSIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROINTESTINAL DYSPLASIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
LARGE INTESTINE PERFORATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 3 | 0 | 1
ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
FURUNCLE (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 3 | 4 | 0 | 3 | 1 | 0
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PELVIC ABSCESS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
VULVAL ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
ACARODERMATITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0 | 0
ABDOMINAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
ABSCESS INTESTINAL (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 0 | 1
URETHRAL CYST (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
PURPURA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
BURNS SECOND DEGREE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
THERAPEUTIC AGENT TOXICITY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
OSTEONECROSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
OSTEOPOROTIC FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0
ASTHENIA (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
CHEST DISCOMFORT (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 0 | 0
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHRONIC LYMPHOCYTIC LEUKAEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABA 30/~10mg/kg (IP) (N=65) | ABA 3mg/kg (IP) (N=130) | ABA ~10mg/kg (IP) (N=128) | ABA ~10mg/kg (MP) (N=44) | ABA ~10mg/kg (OL) (N=324) | Placebo (IP) (N=128) | Placebo (MP) (N=46)
HEADACHE (Nervous system disorders) | 7 | 12 | 13 | 2 | 30 | 8 | 3
DIZZINESS (Nervous system disorders) | 4 | 4 | 3 | 0 | 3 | 3 | 1
NAUSEA (Gastrointestinal disorders) | 6 | 11 | 9 | 5 | 35 | 9 | 2
VOMITING (Gastrointestinal disorders) | 5 | 3 | 2 | 3 | 23 | 8 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 3 | 7 | 3 | 26 | 7 | 3
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 3 | 0 | 0
INFLUENZA (Infections and infestations) | 1 | 2 | 3 | 1 | 13 | 3 | 3
BRONCHITIS (Infections and infestations) | 0 | 1 | 2 | 3 | 6 | 2 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 7 | 2 | 1 | 25 | 5 | 4
URINARY TRACT INFECTION (Infections and infestations) | 1 | 6 | 3 | 1 | 18 | 7 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 5 | 0 | 3 | 25 | 6 | 3
RASH (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 1 | 10 | 2 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7 | 9 | 7 | 3 | 27 | 8 | 3
FATIGUE (General disorders) | 5 | 8 | 4 | 3 | 22 | 10 | 0
PYREXIA (General disorders) | 9 | 4 | 5 | 0 | 21 | 10 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.